CLINICAL TRIAL: NCT01375556
Title: Genetics of the Acute Response to Alcohol in Humans
Brief Title: Genetics of the Acute Response to Alcohol in Social Drinkers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: 110180; 11-AA-0180
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2016-01-20

CONDITIONS: Alcoholism; Genetics
Keywords: Alcohol Clamp; Pharmacogenetics; Family History of Alcoholism; Pharmacodynamics; Healthy Volunteer; HV
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

INTERVENTIONS:
Drug: Ethanol

SUMMARY:
Background:

- Previous research has shown that a person s genes can influence how they respond to alcohol. But researchers do not yet know all the genes that might be involved.

Objectives:

- To identify genes that are related to how non-alcoholic individuals respond to alcohol.

Eligibility:

- Healthy people between 21 and 30 years of age who have no history of alcohol or drug dependence.

Design:

* The study requires one or two 9-hour visits to the National Institutes of Health Clinical Center.
* Participants must not take any medicines (except birth-control pills for women) for at least 3 days before the visit. They must not drink alcohol for at least 2 days before the visit.
* Screening includes a medical history, physical exam, and a urine test for drugs of abuse.
* Participants will be given alcohol over about 2.5 hours. This will have about the same effect as having three to four drinks. Frequent breathalyzer tests will check breath alcohol level during the infusion.
* Before and during the infusion, participants will complete questionnaires about mood and feelings. Other tests will study thinking, balance, judgment, and risk-taking. Blood samples will be collected four times during the infusion.
* Participants will have breakfast at the start of the visit (around 8:00 AM). They will have a snack before the start of the alcohol infusion (around 10:45 AM). Lunch will be served after the alcohol infusion is complete (around 2:20 PM). After the tests, those in the study will have to stay in the Clinical Center until their breath alcohol level falls below 0.02%. This can take up to 2.5 hours. A final blood sample will be drawn at that time. Participants will not be able to drive themselves home after the study visits. Also, they should not take any medicines or operate any machinery for at least 2 hours after leaving NIH.

DETAILED DESCRIPTION:
Previous research, including our prior studies using the alcohol clamp, has shown substantial genetic influences on alcohol pharmacokinetics and pharmacodynamics. While the influence of several individual genes on alcohol pharmacokinetics and pharmacodynamics has been examined, there has not been a comprehensive evaluation of genetic influences on the pharmacokinetics and pharmacodynamics of alcohol in humans.

Objectives: To evaluate the genetic underpinnings of the pharmacodynamics of alcohol using candidate gene analysis of measures of the initial and adaptive acute response to alcohol in humans.

Study Population: Subjects will be 21-30 year-old non-smoking, male and female non-dependent drinkers in good health, as determined by medical history, physical exam, and ECG and lab tests. Subjects with Axis-I psychiatric diagnoses, including alcohol or substance dependence, will be excluded.

Design: The study will be conducted in two phases. In phase I, 40 subjects (20 with positive family history of alcoholism (FHP) and 20 with no family history of alcoholism (FHN)) will undergo two ethanol infusion sessions to compare different breath alcohol concentration exposures. In one session (Clamp session), participants will be infused with 6% ethanol in saline using an individualized infusion profile to achieve and clamp breath alcohol concentrations (BrAC) at 60 mg% for 2 hours. In the other session (Oral-mimic session), participants will be infused with 6% ethanol and saline using another individualized infusion profile to achieve a BrAC-time profile that would be typically obtained after oral administration (ascending limb to peak BrAC followed by descending limb). During each session, serial BrACs will be obtained, and heart-rate and skin blood flow will be continuously recorded. A battery of subjective (self-rating questionnaires) and objective measures (psychomotor performance, behavioral disinhibition tasks) will be obtained at baseline and two points during the infusion to assess the initial response and adaptive response to alcohol. The measures of initial response and adaptive response will be compared between sessions to determine which provides greater sensitivity (higher effect size) for detecting family history differences.

In phase II, 160 participants will undergo a one session study. Participants will receive an ethanol infusion to achieve the BrAC-time profile (Clamp or Oral-mimic) that provides the greater sensitivity to family history of alcoholism in phase I of the study. The same battery of subjective and objective measures will be obtained to assess the initial response and adaptive response to alcohol. These response measures will be used as endophenotypes for examination of genetic association with a set of candidate genes, based on previous clinical and pre-clinical studies.

Outcome measures: Initial response to alcohol and adaptive response to alcohol measures will be obtained for a battery of assessments, including subjective ratings of alcohol effects, psychomotor performance, behavioral disinhibition tasks and autonomic measures.

ELIGIBILITY:
* INCLUSION CRITERIA:

Male and female participants between 21-30 years of age.

Good health as determined by medical history, physical exam, EKG and lab tests.

EXCLUSION CRITERIA:

Current or prior history of any disease, including CNS, cardiovascular, respiratory, gastrointestinal, hepatic, renal, endocrine, or reproductive disorders.

Positive hepatitis or HIV test at screening.

Current (i.e., in the past year) diagnosis of Axis-I psychiatric illness.

Current or lifetime diagnosis of alcohol or substance dependence.

Currently (i.e., in the past year) seeking treatment for alcohol-related problems.

Non-drinkers (alcohol-na(SqrRoot) ve individuals or current abstainers), or individuals who have never consumed more than 4 drinks on at least one occasion.

Current or prior history of alcohol-induced flushing reaction, including rapid reddening of the face, rapid heart rate and breathing, and nausea after 1 or 2 drinks.

Regular tobacco users will be excluded from the study in order to avoid nicotine withdrawal symptoms. Occasional use of tobacco products (up to 20 cigarettes/week, Fagerstrom Test for Nicotine Dependence Score less than 4) is acceptable.

Positive result on urine drug screen or breathalyzer test at screening

No regular use of medications for the last 3 months. Use of prescription or OTC medications known to interact with alcohol within 2 weeks of the study. These include, but may not be limited to: isosorbide, nitroglycerine, benzodiazepines, warfarin, anti-depressants such as amitriptyline, clomipramine and nefazodone, anti-diabetes medications such as glyburide, metformin and tolbutamide, H2-antagonists for heartburn such as cimetidine and ranitidine, muscle relaxants, anti-epileptics including phenytoin and phenobarbital codeine, and narcotics including darvocet, percocet and hydrocodone. Drugs known to inhibit or induce enzymes that metabolize alcohol should not be used for 4 weeks prior to the study. These include chlorzoxazone, isoniazid, metronidazole and disulfiram. Cough-and-cold preparations which contain anti-histamines, pain medicines and anti-inflammatories such as aspirin, ibuprofen, acetaminophen, celecoxib and naproxen, should be withheld for at least 72 hours prior to each study session.

Females must not be pregnant or breast-feeding. Female participants will undergo a urine beta-hCG test to ensure they are not pregnant during screening and study visits.

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2011-05-26; Primary Completion 2016-01-20 (Actual); Study Completion 2016-01-20 (Actual)

PRIMARY OUTCOMES:
Initial response to alcohol and adaptive response to alcohol measures for subjective ratings of alcohol effects, psychomotor performance, behavioral disinhibition tasks and autonomic measures

CONTACTS AND LOCATIONS:
Overall Officials: Vijay A Ramchandani, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bernstein DP, Stein JA, Newcomb MD, Walker E, Pogge D, Ahluvalia T, Stokes J, Handelsman L, Medrano M, Desmond D, Zule W. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child Abuse Negl. 2003 Feb;27(2):169-90. doi: 10.1016/s0145-2134(02)00541-0. PMID 12615092
- [Background] Bierut LJ, Agrawal A, Bucholz KK, Doheny KF, Laurie C, Pugh E, Fisher S, Fox L, Howells W, Bertelsen S, Hinrichs AL, Almasy L, Breslau N, Culverhouse RC, Dick DM, Edenberg HJ, Foroud T, Grucza RA, Hatsukami D, Hesselbrock V, Johnson EO, Kramer J, Krueger RF, Kuperman S, Lynskey M, Mann K, Neuman RJ, Nothen MM, Nurnberger JI Jr, Porjesz B, Ridinger M, Saccone NL, Saccone SF, Schuckit MA, Tischfield JA, Wang JC, Rietschel M, Goate AM, Rice JP; Gene, Environment Association Studies Consortium. A genome-wide association study of alcohol dependence. Proc Natl Acad Sci U S A. 2010 Mar 16;107(11):5082-7. doi: 10.1073/pnas.0911109107. Epub 2010 Mar 2. PMID 20202923
- [Background] Blekher T, Ramchandani VA, Flury L, Foroud T, Kareken D, Yee RD, Li TK, O'Connor S. Saccadic eye movements are associated with a family history of alcoholism at baseline and after exposure to alcohol. Alcohol Clin Exp Res. 2002 Oct;26(10):1568-73. doi: 10.1097/01.ALC.0000033121.05006.EF. PMID 12394291